CLINICAL TRIAL: NCT05330273
Title: A Phase I, Open-label, Fixed-sequence, Two-period, Crossover, Drug-drug Interaction Study to Investigate the Effect of Efavirenz on the Pharmacokinetics of Ganaplacide and Lumefantrine Combination in Healthy Participants
Brief Title: Drug-drug Interaction Study of Ganaplacide and Lumefantrine With Efavirenz
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CKAF156A2107
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Malaria
Keywords: Drug-drug interaction; DDI; ganaplacide; lumefantrine; efavirenz; Pharmacokinetic; PK; safety and tolerability; healthy participants
MeSH Terms: conditions — Malaria | interventions — ganaplacide; Lumefantrine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Period 1: KAF156 + LUM566 / Period 2: KAF156 + LUM566 + Efavirenz (Experimental): Participants enrolled will receive a single oral dose of ganaplacide and lumefantrine combination on Day 1 of Period 1.
  In Period 2, participants will receive an oral dose of efavirenz q.d. in the evening on Days 1 through 24 and a single dose of ganaplacide and lumefantrine combination on the morning of Day 11.
  Interventions: Drug: Ganaplacide; Combination Product: Lumefantrine; Drug: Efavirenz

INTERVENTIONS:
Drug: Ganaplacide — Period 1: 400 mg (4 x 100 mg tablets) for oral administration Period 2: 400 mg (4 x 100 mg tablets) for oral administration
  Other Names: KAF156
Combination Product: Lumefantrine — Period 1: 480 mg (2 x 240 mg sachets) for oral administration Period 2: 480 mg (2 x 240 mg sachets) for oral administration
  Other Names: LUM566
Drug: Efavirenz — Period 2: 600 mg (1 x 600 mg tablet) for oral administration once daily (q.d.)

SUMMARY:
This study assessed the effect of multiple doses of a moderate inducer of cytochrome P450 (CYP) 3A4 (efavirenz) on the pharmacokinetics (PK) of ganaplacide and lumefantrine combination. Results from this study will provide guidance on prescribing ganaplacide and lumefantrine combination when co-administered with moderate inducers of CYP3A4.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence, 2-period, crossover, Drug-drug interaction (DDI) study, to evaluate the effect of multiple doses of efavirenz on the single-dose PK of ganaplacide and lumefantrine in healthy participants. The study consisted of a screening period of up to 28 days, 2 Baseline evaluations (on Day 1 of each treatment period), and 2 treatment periods which were separated by a washout period.

Participants who meet the eligibility criteria at Screening were admitted to the study site for First Baseline evaluations on Day -1 of Period 1. Baseline safety assessments were performed prior to first dosing of study treatment in each period. The participants were domiciled from the First Baseline visit until the end of the PK sampling in Period 1 and were released from the site. Participants returned to the site for the Second Baseline visit and were domiciled until the Study Completion visit in Period 2.

Participants enrolled received a single oral dose of ganaplacide and lumefantrine combination under fasting conditions on Day 1 of Period 1. In Period 2, participants received an oral dose of efavirenz q.d. under fasting conditions in the evening on Days 1 through 24 and a single dose of ganaplacide and lumefantrine combination under fasting conditions on the morning of Day 11. Between the two treatment periods, there was a washout period of at least 14 days, beginning from the last PK sample collection in Period 1 and continuing until the first dose of study treatment in Period 2.

Safety assessments (including physical examinations, ECGs, vital signs, clinical laboratory evaluations, C-SSRS, and AE and SAE monitoring) were performed during the study. The Study Completion evaluations occurred on Day 25 of Period 2, followed by a post-study safety contact (e.g. follow-up telephone call, email) approximately 30 days after the last dose of study treatment. Total duration of study was approximately 55 days from the First Baseline visit to the Study Completion visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Healthy male and non-childbearing potential female participants 18 to 55 years of age inclusive, at Screening.
* In good health as determined by medical history, physical examination, vital signs, ECG and clinical laboratory tests, at Screening.
* Must weigh at least 50 kg with a body mass index (BMI) within the range of 18.0 to 29.9 kg/m2 inclusive, at Screening.

Exclusion Criteria:

* Known family history or presence of long QT syndrome.
* Known history or current clinically significant arrhythmias.
* Any single parameter of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), or alkaline phosphatase (ALP) exceeding 1.2 x upper limit of normal (ULN) and total bilirubin ≥ 1.5 x ULN or any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or serum bilirubin at Screening or First Baseline.
* History of psychiatric illness.
* Score "yes" on item 4 or item 5 of the suicidal ideation section of the C-SSRS, if this ideation occurred in the past 6 months of Screening, or "yes" on any item of the suicidal behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the suicidal behavior section), if this behavior occurred in the past 2 years of Screening.
* History or presence of seizures.
* History or presence of duodenal ulcer, ulcerative colitis or Crohn's disease.
* Presence of active or uncontrolled thyroid disease.

Additional protocol-defined inclusion / exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) to the 24-hour time point (AUC^0-24) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC^0-24 will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Apparent total body clearance of drug from plasma following extravascular administration (CL/F) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL/F will be listed and summarized using descriptive statistics
Apparent volume of distribution during terminal elimination phase following extravascular administration (Vz/F) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz/F will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T^1/2 will be listed and summarized using descriptive statistics.

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) to the 24-hour time point (AUC0-24) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC^0-24 will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T^1/2 will be listed and summarized using descriptive statistics.
Metabolite to Parent Ratio (MR) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. MR will be listed and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided